CLINICAL TRIAL: NCT01572597
Title: Increased Second-line Eradication Rate of Helicobacter Pylori by Adding N-acetylcystein or Metronidazole to the Conventional Triple Therapy.
Brief Title: Increased Re-eradication Rate of Helicobacter Pylori by Adding N-acetylcystein or Metronidazole to the Triple Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Ming-Cheh Chen, Principal Investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB100-26
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
Keywords: Helicobacter pylori; antibiotic resistance; N-acetylcystein; biofilm; second-line eradication treatment
MeSH Terms: interventions — Rabeprazole; Clarithromycin; Acetylcysteine; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylcystein (Experimental): 10-day triple therapy plus N-acetyl-cystein to remove the biofilm.
  Interventions: Drug: 10RAC+acetylcystein
- Metronidazole (Active Comparator): 10-day triple therapy plus metronidazole (concomitant therapy) as active comparator
  Interventions: Drug: 10RAC+metronidazole

INTERVENTIONS:
Drug: 10RAC+acetylcystein — 10-days rabeprazole 20mg b.i.d + clarithromycin 500mg b.i.d + amoxicillin 1000mg b.i.d + N-acetyl-cystein 600mg b.i.d
  Other Names: Pariet; Klaricid; Hiconcil; Fluimucil
  Arms: Acetylcystein
Drug: 10RAC+metronidazole — 10-days rabeprazole 20mg b.i.d + clarithromycin 500mg b.i.d + amoxicillin 1000mg b.i.d + metronidazole 500mg b.i.d
  Other Names: Pariet; Klaricid; Hiconcil; Flagyl
  Arms: Metronidazole

SUMMARY:
Compare efficacy and safety of 10-day triple therapy (rabeprazole, clarithromycin and amoxicillin) plus N-acetylcystein versus 10-day concomitant therapy (rabeprazole, clarithromycin, amoxicillin and metronidazole) for re-eradication for gastric Helicobacter pylori infection.

DETAILED DESCRIPTION:
Background: Antimicrobial resistance has decreased the eradication rates of common used triple therapy for Helicobacter pylori infection (less than 80%). Such treatment for patient previously with treatment failure, the retreatment eradication rate is less then 50%. Some studies showed the Helicobacter pylori form biofilm to prevent entry of antibiotics, and the N-acetylcystein is helpful to dissolve the biofilm.

Objective: To determine the eradication rate of the common used triple therapy after adding N-acetylcystein for second line treatment for adults infected with Helicobacter pylori in Eastern Taiwan.

Design: Randomized, open-label, prospective controlled trial.

Patients: who are previously failed the primary treatment for eradication and still infected by Helicobacter pylori.

Measurements: 13C-urea breath test, upper endoscopy, histologic evaluation, rapid urease test, bacterial culture, assessment of antibiotic resistance and CYP2C19 genotype of host.

Intervention: patients with Helicobacter pylori eradication treatment failure are recruited and randomly assigned to receive one of the following therapeutic schemes: 1) study group: rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + N-acetylcystein 0.6g bid for 10 days; 2) control group: rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for 10 days. Repeat upper endoscopy for histologic evaluation, rapid urease test or 13C-urea breath test after 4 week of treatment to assess the treatment result. The influence on the hybrid therapies of antibiotic resistance of Helicobacter pylori and CYP2C19 genotype of host were determined.

Expected results: The new second line treatment for eradication of Helicobacter pylori is effective, and to determine the relation of antibiotic resistance of Helicobacter pylori and CYP2C19 genotype of host to the treatment result.

ELIGIBILITY:
Inclusion Criteria:

* Patient after treatment for Helicobacter pylori eradication.
* Still clinically with evidence of gastric Helicobacter pylori infection.

Exclusion Criteria:

* woman in breast feeding or pregnancy.
* allergy to drugs used in study.
* never treated for H. pylori.
* intolerance to fructose, lactose.
* patients with hematologic, brain or spinal disorders.
* patients under 20 years old.
* patients with malignancy or with decompensated function of vital organs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Re-eradication rate | 4 weeks after complete use of drug for treatment
  A negative post-treatment 13C-urea breath test result at more than 4 weeks after complete use of drug for treatment.

SECONDARY OUTCOMES:
Influence of Participant's CYP2C19 genotype on re-eradication rate | 4 weeks after complete use of drug for treatment
  Influence of Participant's CYP2C19 genotype (EM, IM or PM) on re-eradication rate of Helicobacter pylori

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheh CHEN, MD, Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan, Taiwan

REFERENCES:
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Cammarota G, Branca G, Ardito F, Sanguinetti M, Ianiro G, Cianci R, Torelli R, Masala G, Gasbarrini A, Fadda G, Landolfi R, Gasbarrini G. Biofilm demolition and antibiotic treatment to eradicate resistant Helicobacter pylori: a clinical trial. Clin Gastroenterol Hepatol. 2010 Sep;8(9):817-820.e3. doi: 10.1016/j.cgh.2010.05.006. Epub 2010 May 31. PMID 20478402